CLINICAL TRIAL: NCT07387783
Title: The Association Between Sleep Quality and Cognitive Functions in Healthy Young Adults
Brief Title: Sleep Quality and Cognitive Functions in Adults: A Cross-Sectional Study
Status: Not yet recruiting | Type: Observational
Sponsor: Uskudar University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Fatma Demir, Principal Investigator, Uskudar University
Other Study IDs: 61351342/020-1143; TUBITAK 2209A 1919B012466805 (Other Grant/Funding Number: The Scientific and Technological Research Council of Turkey (TUBITAK))
Record Dates: First submitted 2026-01-21; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Sleep Quality; Cognitive Functions
Keywords: sleep quality; Cognitive Function; Young Adults; verbal memory; wearable device
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Young Adults: Healthy young adult participants without diagnosed neurological, psychiatric, or sleep disorders who undergo assessment of sleep quality and cognitive functions during a single observational assessment period.

SUMMARY:
This observational cross-sectional study aims to examine the association between sleep quality and cognitive functions in healthy young adults. Subjective sleep quality will be assessed using the Pittsburgh Sleep Quality Index, and objective sleep parameters will be collected using a wearable device over five consecutive days. Cognitive functions will be evaluated at a single assessment session using standardized neuropsychological tests, including measures of attention, executive functions, and verbal memory. The study seeks to explore relationships between subjective and objective sleep measures and cognitive performance. Findings from this study may contribute to a better understanding of how sleep quality is associated with cognitive functioning in healthy young adults.

DETAILED DESCRIPTION:
This study is designed as an observational, cross-sectional investigation conducted in healthy young adults to examine the association between sleep quality and cognitive functions. Participants will be recruited from a non-clinical population and will undergo a single assessment period. Subjective sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), a self-report questionnaire evaluating sleep quality and sleep-related disturbances over the previous month. In addition to subjective measures, objective sleep parameters will be collected using a wearable device worn continuously for five consecutive days. Wearable-derived sleep metrics will include total sleep time, sleep efficiency, sleep onset latency, and wake after sleep onset, as provided by the device's standard algorithms. Cognitive functions will be evaluated during a single in-person assessment session following completion of the sleep data collection period. Cognitive assessment will include standardized neuropsychological tests measuring attention, executive functions, and verbal memory. Attention and executive functions will be assessed using the Victoria Stroop Test, and verbal memory processes will be evaluated using the Öktem Verbal Memory Processes Test, administered according to standardized procedures. Demographic information and relevant background variables will be collected to characterize the study sample. Statistical analyses will primarily focus on examining associations between subjective and objective sleep parameters and cognitive test outcomes. Correlation analyses and multivariable statistical models may be used to explore relationships between sleep quality and cognitive performance while accounting for potential confounding variables. This study aims to contribute to the understanding of how variations in sleep quality are associated with cognitive functioning in healthy young adults, using both subjective and objective sleep measures.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 35 years.
* Ability and willingness to provide written informed consent.
* Sufficient ability to read, understand, and communicate in Turkish, the language in which the assessments are administered.
* Self-reported good general health, with no active medical or psychiatric conditions that significantly affect daily functioning.
* Willingness and ability to wear a wearable sleep monitoring device continuously for five consecutive days and to comply with device usage instructions.
* Ability to attend and complete a single-session cognitive assessment

Exclusion Criteria:

* Regular or frequent use of medications known to affect sleep or cognitive function, including sedative-hypnotics, benzodiazepines, antipsychotics, stimulants, opioids, or similar agents.
* Initiation of, or dose changes in, psychotropic medications within the past four weeks.
* Being under the influence of alcohol or illicit substances on the day of cognitive testing.
* Engagement in night shift work or rotating shift schedules within the past one month.
* Travel across time zones resulting in a time difference of two hours or more within the past two weeks.
* Uncontrolled high daily intake of caffeine (e.g., >400 mg/day) and unwillingness to reduce consumption during the study period.
* Color blindness or other color vision deficiencies, due to their potential impact on Stroop Test performance.
* Dermatological conditions, allergies, or skin lesions at the wrist that prevent wearing the device, or refusal to wear the device as required.
* Acute illness within the past two weeks, including febrile infections, severe pain, or other acute medical conditions that may temporarily affect sleep or cognitive performance.
* Pregnancy or early postpartum period.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of healthy young adults aged between 18 and 35 years. Participants are recruited from a non-clinical population and are required to be fluent in Turkish to ensure valid administration of cognitive assessments. Individuals with self-reported good general health and without active medical, neurological, or psychiatric conditions that may affect sleep or cognitive functioning are eligible. All participants are able and willing to comply with the study procedures, including wearing a wearable sleep monitoring device for five consecutive days and completing a single-session cognitive assessment.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Composite Objective Sleep Quality Index Derived From Wearable Device | During 5 consecutive days around baseline assessment
  A composite objective sleep quality index will be derived from wearable device data collected continuously over five consecutive days. The composite score will be calculated by combining standardized values of total sleep time, sleep efficiency, sleep onset latency, and wake after sleep onset into a single summary measure representing overall objective sleep quality.

SECONDARY OUTCOMES:
Sleep Quality (Pittsburgh Sleep Quality Index Scores) | Baseline (single assessment)
  Subjective sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The total PSQI score ranges from 0 to 21, with higher scores indicating poorer sleep quality.
Cognitive Performance (Victoria Stroop Test Scores) | Baseline (single assessment)
  Attention and executive functions will be assessed using the Victoria Stroop Test. Outcome measures include completion time and error scores obtained during the test.
Verbal Memory Performance (Öktem Verbal Memory Processes Test Scores) | Baseline (single assessment)
  Verbal memory will be evaluated using the Öktem Verbal Memory Processes Test. Outcome measures include standardized scores reflecting learning and recall performance.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Demir, MSc, Principal Investigator — Üsküdar University
Locations (1):
- Üsküdar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves sensitive personal data related to sleep patterns and cognitive performance, and participant consent for data sharing was not obtained. Data will be used solely for the purposes defined in the approved study protocol.